CLINICAL TRIAL: NCT06786494
Title: Tart Cherry Juice for Sleep in Older Adults With Insomnia: A Pilot Study of Feasibility and Comprehensive Mechanisms
Acronym: CherryZZZ
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Courtney Millar (Other)
Responsible Party: Sponsor-Investigator, Courtney Millar, Assistant Scientist II, Hebrew SeniorLife
Organization: Hebrew SeniorLife (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: CherryZZZ
Record Dates: First submitted 2025-01-10; First posted 2025-01-22 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Sleep Problems; Insomnia
Keywords: Montmorency; cherry; flavonoids; sleep quality
MeSH Terms: conditions — Parasomnias; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tart Cherry Juice (Experimental)
  Interventions: Other: Tart Cherry Juice
- Placebo Juice (Placebo Comparator)
  Interventions: Other: Placebo juice

INTERVENTIONS:
Other: Tart Cherry Juice — Individuals will be asked to consume 240 mL (i.e., 8 ounces) at approximately 5 pm and 240 mL (i.e., 8 ounces) of tart cherry juice at approximately 1 hour before bedtime for 4 weeks.
  Arms: Tart Cherry Juice
Other: Placebo juice — Individuals will be asked to consume 240 mL (i.e., 8 ounces) at approximately 5 pm and 240 mL (i.e., 8 ounces) of placebo juice at approximately 1 hour before bedtime for 4 weeks.
  Arms: Placebo Juice

SUMMARY:
The purpose of this research study is test if a study that asks older adults with sleep problems to consume tart cherry products is feasible and determine if it can change sleep patterns. This study is a total of 12 weeks. Participants will be asked to consume tart cherry juice for 4 weeks and the placebo juice for 4 weeks, while wearing a digital monitor that measures sleep. Blood (about 3 teaspoons) and urine (about 2 tablespoons) samples will be taken before and after consuming both juices to measure certain biological markers related to sleep.

DETAILED DESCRIPTION:
The overall goal of this study is to determine feasibility of a tart cherry juice intervention in older adults, and generate preliminary data of outcomes and mechanisms related to sleep. We propose a 2-arm randomized, double-blind, cross-over study in 20 older adults with self-reported insomnia. Participants will consume 240 mL of tart cherry juice or placebo (calorically matched to the tart cherry juice beverage, but theoretically devoid of melatonin, tryptophan, magnesium and flavonoids), twice/evening for 4 weeks in a randomly assigned order.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged ≥65 years
* Self-reporting insomnia (e.g., trouble sleeping approximately 3 nights a week for at least 6 months and/or an Insomnia Severity Index score ≥ 10 points)
* Usual bed-time between 8:00 pm and 1:00 am

Exclusion Criteria:

* Unwilling to follow the study protocol
* Inability to properly use the wearable device, complete smartphone-based surveys, or follow the intervention protocol
* Self-report of medically diagnosed sleep disorders except insomnia (e.g., sleep apnea)
* Current and consistent use of sleep aids or hypnotic prescriptions (e.g., trazadone)
* Self-report of cognitive impairment, dementia, or other neurological disorder
* Are on unstable medications (i.e., change within the last 3 months) for other conditions
* Have an allergy to the intervention products
* Self-report history of diabetes
* Current alcohol (Alcohol Use Disorders Identification Test ≥4 points33,34) or drug use disorder (Drug Abuse Screening Test,35,36 DAST-10>2 points)
* Are excessive caffeine drinkers (>5 cups of caffeinated beverages a day)
* Any other reason/condition the PI and investigative team believe this intervention would be unsafe

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 20 (Actual)
Dates: Start 2025-01-15 (Actual); Primary Completion 2025-08-13 (Actual); Study Completion 2025-08-13 (Actual)

PRIMARY OUTCOMES:
Recruitment Rate | From first contact until randomization
  Number of individuals that need to be screened to be enrolled that are randomized to the intervention.
Attrition | From randomization until end of 12 week study
  Number of individuals randomized that withdraw from the intervention after randomization and starting the intervention product.
Compliance | From randomization until end of 12 week study
  The number of doses consumed/ the number of intended doses (%)
Ability to Collect Data | From enrollment to end of 12 week study
  The percentage of missing data points from electronic capture data devices.
Practicality | Week 12 study visit
  Self-reported willingness to continue the dietary regimen after study completion.

SECONDARY OUTCOMES:
Sleep Quantity (minutes) | From enrollment to end of 12 week study
Sleep Quality | Week 1, Week 5, Week 8, Week 12
  The validated self-report questionnaire, the Pittsburg Sleep Quality Index, will be used as a measure of sleep quality. This instrument ranges from 0-21 points, with higher scores indicating worse sleep quality.
Urinary melatonin metabolite (6-sulphatoxymelatonin) | Week 1, Week 5, Week 8, Week 12
Serum Marker of Serotonin (kynurenine/tryptophan ratio in blood) | Week 1, Week 5, Week 8, Week 12
Urinary Cortisol | Week 1, Week 5, Week 8, Week 12
Interleukin 6 in blood | Week 1, Week 5, Week 8, Week 12
C-reactive Protein in Blood | Week 1, Week 5, Week 8, Week 12

OTHER OUTCOMES:
Mood | Week 1, Week 3, Week 5, Week 8, Week 10, Week 12
  A validated self-report questionnaire, the Center for Epidemiological Studies Depression Scale, will be used to evaluate mood/depressive symptom severity. This instrument ranges from 0-60 points, with higher scores indicating more severe symptoms of depression.
Stress | Week 1, Week 3, Week 5, Week 8, Week 10, Week 12
  The validated self-report questionnaire, the Perceived Stress Scale, will be used to evaluate stress. This instrument ranges from 0-56 points, with higher scores indicating more stress.
Pain | Week 1, Week 3, Week 5, Week 8, Week 10, Week 12
  The validated self-report questionnaire, the Geriatric Pain Measure, will be used to evaluate pain. This instrument ranges from 0-42 points, with higher scores indicating more severity of pain.

CONTACTS AND LOCATIONS:
Overall Officials: Courtney Millar, PhD, Principal Investigator — Hebrew SeniorLife, Marcus Institute of Aging, Harvard Medical School
Locations (1):
- Hebrew Rehabilitation Center, Roslindale, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided